CLINICAL TRIAL: NCT04479085
Title: The Effect of Nursing Initiative for Home Environment Regulation on Symptom Control and Quality of Life in Children With Allergic Rhinitis: A Randomized Controlled Study
Brief Title: Effect of Home Environment Regulation on Symptom Control and Quality of Life in Children With Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, muradiye aldem budak, research assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: maldem
Record Dates: First submitted 2020-07-06; First posted 2020-07-21 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; children; nursing; Allergic Rhinitis Due to House Dust Mite
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Methods

STUDY DESIGN:
Intervention Model Description: pretest-posttest, parallel group, randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The nursing attempt to organize the home environment for the experimental group will take 17 weeks. During this period, two home visits and two telephone calls will be made. During the first home visit, training will be organized to regulate the home environment. Temperature and humidity changes of the houses will be monitored during the operation with the heat-moisture meter device. Children in this group will be given an anti-allergic duvet cover. Home environment arrangements of mothers and changes in the quality of life of children will be examined at the beginning and end of the study. Children's symptoms will be monitored weekly for 17 weeks.
  Interventions: Other: nursing intervention
- control group (No Intervention): No intervention will be made on the control group. The humidity and temperature changes in the home environment of the children in this group and their symptoms will be monitored on a weekly basis during the study.

INTERVENTIONS:
Other: nursing intervention — It includes individual trainings for the regulation of the home environment,
  give a booklet
  to reinforce education and to give anti-allergic bedding sets.
  Arms: experimental group

SUMMARY:
The purpose of this study is to examine the effect of nursing intervention to regulate the home environment on symptom control and quality of life in children with allergic rhinitis.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a clinical picture resulting from one or more allergen sensitivities. Seasonal AR develops due to grass, tree and grass pollen. Prennial AR develops due to house dust mite, cockroaches, mold and pets.The prevalence of allergic rhinitis in children ranges from 19.3-50.8%. AR affects school performance, sleep patterns and quality of life in children.Children spend most of their lives in the home environment, and many studies have shown that AR is associated with the home environment in children. Control measures should be taken in patients' homes to prevent and reduce the symptoms of allergic rhinitis in children. Awareness and education should be provided to families and children about the importance of these measures.

This study is a pretest-posttest, parelel group, randomized controlled study study to examine the effect of nursing intervention to regulate the home environment on symptom control and quality of life in children with allergic rhinitis.

sample of the study; The effect size was intended to be medium effect size due to the absence of a similar randomized controlled study to determine the quality of life in children with allergic rhinitis. In the study, the number of samples to be included in the study with 0.7 medium effect size, power 80%, alpha reliability level 95%, 26 experiments and 26 controls were calculated as 52 children and their mothers.

Randomized appointments were made in the appointment of 52 children and mothers who were followed up with the diagnosis of allergic rhinitis, who included the criteria for inclusion and exclusion, and who volunteered to participate in the study. Stratified randomization method was used in this study. Stratified randomization method was used in this study. The gender of the children (girls and boys), the age of the children (6-9 years, 10-12 years) and the level of mother education (primary education, high school, university) were determined as prognastic factors for stratification. Randomization was performed in a total of 52 participants, 26 experimental and 26 control groups.

Number, percentage, average and standard deviation will be used in the evaluation of the descriptive data obtained from the research; Significance will be evaluated within 95% confidence interval, p <0.05 will be taken.

The nursing attempt to organize the home environment for the experimental group will take 17 weeks. During this period, two home visits and two telephone calls will be made. During the first home visit, training will be organized to regulate the home environment, as well as a heat-moisture meter and anti-allergic duvet cover set.

There will be two home visits to the control group. During the first home visit, a heat-humidity meter device will be given. Data collection forms will be applied at the beginning and end of the study.training will be organized at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The child is diagnosed with allergic rhinitis
* 6-12 age group children
* The child's sensitivity to at least one of Dermatophagoides pteronyssinus and/or Dermatophagoides farinae according to the skin prick test.
* Although sensitive to at least one of the house dust mites Dermatophagoides pteronyssinus and/or Dermatophagoides farinae according to the child's skin pric test;

  * The child has mold allergy according to the skin prick test
  * The child is allergic to cockroaches according to the skin prick test
  * The child has any of the cat and dog allergies according to the skin prick test
* Volunteering to participate in the research

Exclusion Criteria:

* The child has an additional chronic disease other than allergic rhinitis
* Pol The child is allergic to pollen according to the skin prick test
* Child and mother are not literate in Turkish Communication barriers in children and mothers (seeing, hearing, diagnosed mental and mental problems)
* Lack of up-to-date family phone information
* Child and mother living outside the city center

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire for 6-12 Years Old Children with Allergy in the Nose and Eyes (pediatric rinitis quality of life questionnaire PRQLQ) | It will be monitored at the beginning and end of the study.
  Average quality of life score of children will be taken by using the Quality of Life Survey for 6-12 Years Old Children with Allergy in their Nose and Eyes. The scale includes scoring between 0-6 High average score indicates low quality of life.

SECONDARY OUTCOMES:
home environment regulation | It will be monitored at the beginning and end of the study.
  The average score will be taken using the home environment evaluation form.this form was created by researchers.
symptom monitoring | It will be monitored every week for 17 weeks.
  The form created by the researchers aims to identify the symptoms of allergic rhinitis.forms are scored between 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Muradiye ALDEM BUDAK, Principal Investigator — Necmettin Erbakan University; Emine GEÇKİL, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan Universty, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No